CLINICAL TRIAL: NCT00110318
Title: A Pragmatic, Randomised Controlled Trial of Physiotherapy and Corticosteroid Injections in Lateral Epicondylalgia
Brief Title: Trial of Physiotherapy and Corticosteroid Injections in Lateral Epicondylalgia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Queensland (Other)
Collaborators: National Health and Medical Research Council, Australia (Other)
Responsible Party: Principal Investigator, Dr Bill Vicenzino, Chair of Sports Physiotherapy, The University of Queensland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H/355/PHYSIO/01/NHMRC; NHMRC#252710
Record Dates: First submitted 2005-05-05; First posted 2005-05-06 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Tennis Elbow; Musculoskeletal Diseases
Keywords: Tennis Elbow; Physical Therapy Techniques; Evidence-Based Medicine; Primary Health Care
MeSH Terms: conditions — Tennis Elbow; Musculoskeletal Diseases | interventions — Musculoskeletal Manipulations; Exercise Therapy

INTERVENTIONS:
Procedure: Manual therapy and therapeutic exercise
Procedure: Corticosteroid injections

SUMMARY:
This randomised controlled trial will evaluate the role of manual therapy and therapeutic exercise and corticosteroid injections in the treatment of lateral epicondylalgia (tennis elbow).

DETAILED DESCRIPTION:
Musculoskeletal conditions account for the third leading cause of health systems expenditure in Australia. Lateral epicondylalgia (tennis elbow) is a painful musculoskeletal condition that is often treated in primary care. Seven out of every 1000 patients seeing their general medical practitioner do so for this condition, though most are not tennis related. On average 10-30% of sufferers take 12 weeks of absenteeism from work and the condition may last 6-48 months.

Two popular treatment options that are commonly prescribed for the management of lateral epicondylalgia are manual therapy/therapeutic exercise and corticosteroid injections. To date there is little evidence that supports manual therapy/therapeutic exercise. This lack of evidence is largely due to the small number of studies of physiotherapy treatments, most of which are of poor quality. The small number of studies of manual therapy contrasts with the larger number of studies of corticosteroid injections, which show that corticosteroid injections are beneficial in the short term (3-6 weeks), but they are associated with significantly greater recurrence rates and offer no advantage in the long term (12 months). The efficacy of a manual therapy and therapeutic exercise programme compared to that of corticosteroid injections is unknown at this stage.

This randomised controlled trial will evaluate the role of manual therapy and therapeutic exercise in the treatment of lateral epicondylalgia. The factors associated with success or failure of these common treatment options for lateral epicondylalgia will also be examined. A tangible outcome of this project will be the development of clinical guidelines for the most effective method of treating lateral epicondylalgia.

ELIGIBILITY:
Inclusion Criteria:

* Elbow pain for at least 6 weeks and satisfy the widely accepted diagnostic criteria of lateral epicondylalgia
* Diagnostic criteria are pain over the lateral humeral epicondyle that is provoked by gripping activities
* Reduced grip strength and increased sensitivity to manual palpation over the lateral epicondyle
* Reproduction of pain with stretching of the forearm extensor muscles or with specific resisted static contraction of extensor carpi radialis brevis is also usually present.

Exclusion Criteria.

* In the preceding 6 months, had consulted a health care practitioner for neck or arm pain or injury, other than lateral epicondylalgia, which has prevented participation in usual work or recreational activities
* Had treatment with physiotherapy or corticosteroid injections for lateral epicondylalgia in the preceding 6 months
* Upper limb fractures
* Diseases of the bone, muscle and nervous systems that preclude treatment by any of the treatments being evaluated in the project.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198
Dates: Start 2002-03; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
General improvement
Assessors assessment of severity
Pain free grip strength

SECONDARY OUTCOMES:
Global perceived effect score
Pain Visual Analogue Scale
Function Visual Analogue Scale
Impact on occupational and recreational activities
Stratford pain free function questionnaire
Patient rated evaluation questionnaire
Pressure pain threshold
Maximum grip strength
Pain visual analogue scale with gripping
Tests of motor control (reaction time, speed, accuracy, coordination)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Bill Vicenzino, PhD, Principal Investigator — The University of Queensland
Locations (1):
- Musculoskeletal Pain & Injury Research Unit, Division of Physiotherapy, The University of Queensland, Brisbane, Queensland, Australia

REFERENCES:
- [Background] Assendelft WJ, Hay EM, Adshead R, Bouter LM. Corticosteroid injections for lateral epicondylitis: a systematic overview. Br J Gen Pract. 1996 Apr;46(405):209-16. PMID 8703521
- [Background] Mathers C, Penm R. Health systems costs of injury, poisoning and musculskeletal disorders in Australia 1993-94. Australian Institute of Health and Welfare (Health and Welfare Expenditure Series no. 6): Canberra. p 77, 1999.
- [Background] Labelle H, Guibert R, Joncas J, Newman N, Fallaha M, Rivard CH. Lack of scientific evidence for the treatment of lateral epicondylitis of the elbow. An attempted meta-analysis. J Bone Joint Surg Br. 1992 Sep;74(5):646-51. doi: 10.1302/0301-620X.74B5.1388172.
- [Background] Hay EM, Paterson SM, Lewis M, Hosie G, Croft P. Pragmatic randomised controlled trial of local corticosteroid injection and naproxen for treatment of lateral epicondylitis of elbow in primary care. BMJ. 1999 Oct 9;319(7215):964-8. doi: 10.1136/bmj.319.7215.964. PMID 10514160